CLINICAL TRIAL: NCT05877105
Title: Effect of Selected Evidence-based Practices and Related Nurses' Education on the Incidence and Severity of Ventilator-associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, lecturer, Cairo University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NHTMRI-13/23
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Evidence-based Practices; Nursing Education; Incidence; Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: certain VAP bundle as an evidence-based practice will be implemented as the intervention also the needed related nursing education will be given to ensure that the intervention will be implemented properly, and we will examine its effect on VAP incidence and severity among the intervention group as a dependent variable; then, we will compare the finding against the comparative no intervention group who receives the traditional care. Two arms (intervention and non-intervention comparative groups)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-experimental (No Intervention): assessment of MV patients for VAP incidence and severity ICU staff for will be assessed for Compliance with implementing VAP prevention EBP
- experimental (Experimental): The intervention group of patients will receive the proposed VAP prevention EBP which consists of ten items bundle.
  also, assessment of MV patients for VAP incidence and severity ICU staff for will be assessed for Compliance with implementing VAP prevention EBP
  Interventions: Other: Ventilator-associated pneumonia prevention Evidence-based practices (VAPPEBP) which consists of ten items bundle

INTERVENTIONS:
Other: Ventilator-associated pneumonia prevention Evidence-based practices (VAPPEBP) which consists of ten items bundle — VAP prevention EBP which consists of ten items bundle; hand hygiene, head-of-bed elevation, oral care with cetylpyridinium chloride, avoidance of oversedation, proper breathing circuit management, appropriate maintenance of endotracheal tube cuff pressure, closed system and subglottic suctioning, daily assessment for extubation, early ambulation and rehabilitation, and peptic ulcer and deep vein thrombosis (DVT) prophylaxis.
  Arms: experimental

SUMMARY:
Background:

Invasive mechanical ventilation (MV) is used as a cornerstone in the treatment plan of intensive care units (ICUs) patients to provide adequate tissue oxygenation to support the body during the treatment course.

Ventilator-associated pneumonia (VAP) is a preventable iatrogenic complication that can develop in patients undergoing mechanical ventilation. VAP is pneumonia that develops 2 days after endotracheal intubation; the patient must have new or progressive radiological infiltrate, infection alerts (e.g. fever, white blood cell count change), altered sputum characters, and isolation of a causative organism, all together to diagnose VAP. VAP is the most frequent hospital-acquired infection occurring in the ICUs and has a high associated mortality rate. Mortality rate for VAP ranges from 24-51%.

Therefore, this study aims to evaluate the VAP preventive effect of the selected EPB and related nurses' education on the incidence and severity of VAP, as well as assess the nurses' compliance with the selected VAP preventive EBP

Hypothesis:

H1: Implementation of VAP prevention EBP and related nurses' education would reduce the incidence of VAP among mechanically ventilated patients compared to those receiving conventional care.

H2: Implementation of VAP prevention EBP and related nurses' education would reduce the severity of VAP among mechanically ventilated patients compared to those receiving conventional care.

Research question:

Q1: What level of compliance do ICU staff have with implementing of VAP prevention EBP?

Trial design The current study will utilize a prospective, longitudinal, single-arm design, pre & post-experimental. The research's purpose, risks, and potential benefits will be explained to all participants before their voluntary consent and recruitment into the study. Participation was completely voluntary, and written informed consent was obtained from all participants or their families.

ICU nurses will receive tutorial sessions, including four hours of theory and six hours of clinical training in the clinical setting. The tutorial sessions will cover the proper implementation of ten VAP preventive bundles as an EVB. The clinical training will use a demonstration and redemonstration approach to learning to ensure that they understand and can implement the ten VAP preventive bundles efficiently.

Participants sample and setting The study will be held at the ICU of the National Hepatology and Tropical Medicine Research Institute (Imbaba Fever Hospital) (NHTMRI-IFH), Giza, Egypt. The total capacity of the ICUs is 20 beds.

Data collection procedure After obtaining ethical and administrative approval, informed consent will be obtained from eligible patients. The pre-experimental phase will be started by assessing VAP incidence and severity among the participating MV patients using tools 1 and 2, as well as ICU staff compliance to implement the VAP preventive bundle utilizing tool 3 as baseline data for 30-40 days. After finishing the pre-assessment, the following week will be considered washing time before starting the post-experimental time to ensure that all pre-assessment patients are discharged. During the washing time, the nurses will receive a tutorial session on how to implement the adopted VAP preventive bundle, and then the medical and nursing staff will start implementing the VAP preventive bundle in the post-experimental phase for 30-40 days. Tools 1, 2, and 3 will be utilized to evaluate VAP incidence, severity, and ICU staff compliance to implement the VAP preventive bundle. All data will be collected in an Excel sheet for potential statistical analysis.

DETAILED DESCRIPTION:
Background:

Invasive mechanical ventilation (MV) is used as a cornerstone in the treatment plan of intensive care units (ICUs) patients to provide adequate tissue oxygenation to support the body during the treatment course.

Ventilator-associated pneumonia (VAP) is a preventable iatrogenic complication that can develop in patients undergoing mechanical ventilation. VAP is pneumonia that develops 2 days after endotracheal intubation; the patient must have new or progressive radiological infiltrate, infection alerts (e.g. fever, white blood cell count change), altered sputum characters, and isolation of a causative organism, all together to diagnose VAP. VAP is the most frequent hospital-acquired infection occurring in the ICUs and has a high associated mortality rate. Mortality rate for VAP ranges from 24-51%.

Therefore, this study aims to evaluate the VAP preventive effect of the selected EPB and related nurses' education on the incidence and severity of VAP, as well as assess the nurses' compliance with the selected VAP preventive EBP

Hypothesis:

H1: Implementation of VAP prevention EBP and related nurses' education would reduce the incidence of VAP among mechanically ventilated patients compared to those receiving conventional care.

H2: Implementation of VAP prevention EBP and related nurses' education would reduce the severity of VAP among mechanically ventilated patients compared to those receiving conventional care.

Research question:

Q1: What level of compliance do ICU staff have with implementing of VAP prevention EBP?

Trial design The current study will utilize a prospective, longitudinal, single-arm design, pre & post-experimental. The research's purpose, risks, and potential benefits will be explained to all participants before their voluntary consent and recruitment into the study. Participation was completely voluntary, and written informed consent was obtained from all participants or their families.

ICU nurses will receive tutorial sessions, including four hours of theory and six hours of clinical training in the clinical setting. The tutorial sessions will cover the proper implementation of ten VAP preventive bundles as an EVB. The clinical training will use a demonstration and redemonstration approach to learning to ensure that they understand and can implement the ten VAP preventive bundles efficiently.

Participants sample and setting The study will be held at the ICU of the National Hepatology and Tropical Medicine Research Institute (Imbaba Fever Hospital) (NHTMRI-IFH), Giza, Egypt. The total capacity of the ICUs is 20 beds.

Regards to the ICU patients, 72 patients estimated by G power software V.3.1.9.4 (Psychonomic Society, Madison, Wisconsin, USA) with α = 0.05, power (1-β err prob) = 0.80, and effect size = 0.6. Also, eight participants will be added as anticipated dropout during the time of data collection. Hence the total targeted sample size will be 80 patients (40 in each group). Also, all ICU staff (nurses and doctors) working in the selected ICU will be invited to participate in this study to learn and implement the ten VAP preventive bundles.

Data collection procedure After obtaining ethical and administrative approval, informed consent will be obtained from eligible patients. The pre-experimental phase will be started by assessing VAP incidence and severity among the participating MV patients using tools 1 and 2, as well as ICU staff compliance to implement the VAP preventive bundle utilizing tool 3 as baseline data for 30-40 days. After finishing the pre-assessment, the following week will be considered washing time before starting the post-experimental time to ensure that all pre-assessment patients are discharged. During the washing time, the nurses will receive a tutorial session on how to implement the adopted VAP preventive bundle, and then the medical and nursing staff will start implementing the VAP preventive bundle in the post-experimental phase for 30-40 days. Tools 1, 2, and 3 will be utilized to evaluate VAP incidence, severity, and ICU staff compliance to implement the VAP preventive bundle. All data will be collected in an Excel sheet for potential statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients intubated mechanical ventilation for more than 48 hours

Also, the ICU staff (medical or nurses) working in the selected ICU will be invited to participate in this study to learn and implement the ten VAP preventive bundles.

Exclusion Criteria:

* Patients intubated outside the IFH.
* patients have immunocompromised diseases will be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of the selected EPB and related nurses' education on the incidence VAP | 35-40 days
  VAP incidence will be measured using the diagnostic criteria for clinically defined pneumonia outlined by the Centres for Disease Control and Prevention of the United States (TOOL 1) [3]. The ICU specialist will made a final diagnosis of VAP based on chest imaging test results, clinical signs/symptoms, and laboratory findings. VAP incidence will be measured every day for MV patients using tool 1.

SECONDARY OUTCOMES:
Evaluate the effect of the selected EPB and related nurses' education on the severity of VAP | 35-40 days
  The severity of VAP will be determined by sequential organ failure assessment (SOFA) scores [9]. During a patient's stay in the intensive care unit (ICU), the SOFA scoring system employs six reproducible variables per organ system to assess the disease's severity. Vincent et al. developed it in 1996 [9]. Each organ system was assigned a score between 0 (normal) and 4 (most abnormal), with a minimum of 0 and a maximum of 24. We will evaluate the SOFA scores for the patients on ICU admission, the first day of MV connection, every day of VAP development, and on ICU discharge (if applicable).
Assess the compliance of ICU staff with implementing VAP prevention bundel as an EBP | 35-40 days
  VAPPCC is an advanced tool formulated by researchers in terms of the proposed VAP prevention EBP (ten bundle). VAPPCC consists of ten items, including the satisfactory criteria for each item. The ICU staff's compliance for each item ranged from 1 (yes) to 0 (no), with a minimum score of 0 and a maximum of 10. The charge nurse will use VAPPCC to assess the provided care for MV patients daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No